CLINICAL TRIAL: NCT05620355
Title: A Phase 3, Multicentre, Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy and Safety of Daily Oral Administration of BG2109 Alone and in Combination With Add-back Therapy for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women.
Brief Title: Efficacy and Safety of BG2109 in Subjects With Heavy Menstrual Bleeding Associated With Uterine Fibroids.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bio Genuine (Shanghai) Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BG2109-301
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Uterine Fibroids; Heavy Menstrual Bleeding
MeSH Terms: conditions — Leiomyoma; Menorrhagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BG2109 100mg group (Experimental): One tablet of BG2109 100mg + one tablet of placebo for BG2109 + one tablet of placebo for add-back therapy, oral, once-daily.
  Interventions: Drug: BG2109; Drug: Placebo for BG2109; Drug: Placebo for add-back therapy
- BG2109 200mg+ABT group (Experimental): Two tablets of BG2109 100mg + one tablet of add-back therapy, oral, once-daily.
  Interventions: Drug: BG2109; Drug: Add-back therapy
- Placebo group (Placebo Comparator): Two tablets of placebo for BG2109 + one tablet of placebo for add-back therapy, oral, once-daily.
  Interventions: Drug: Placebo for BG2109; Drug: Placebo for add-back therapy

INTERVENTIONS:
Drug: BG2109 — BG2109 100mg film coated tablet for oral administration once daily.
  Arms: BG2109 100mg group; BG2109 200mg+ABT group
Drug: Placebo for BG2109 — Placebo for BG2109 100mg tablet for oral administration once daily.
  Arms: BG2109 100mg group; Placebo group
Drug: Placebo for add-back therapy — Placebo for add-back therapy tablet for oral administration once daily.
  Arms: BG2109 100mg group; Placebo group
Drug: Add-back therapy — Estradiol 1 mg / Norethindrone Acetate 0.5 mg for oral administration once daily.
  Arms: BG2109 200mg+ABT group

SUMMARY:
The primary objective of this study is to demonstrate the superior efficacy versus placebo of BG2109 alone and in combination with add-back therapy for the reduction of heavy menstrual bleeding associated with uterine fibroids in premenopausal women.

DETAILED DESCRIPTION:
The study is a prospective, randomized, parallel group, double-blind, placebo-controlled phase 3 study investigating the efficacy and safety of BG2109 alone and in combination with add-back therapy (Estradiol 1 mg / Norethindrone Acetate 0.5 mg) for the treatment of uterine fibroids in China.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is an 18 years and older premenopausal woman.
2. Subject's Body Mass Index ≥ 18 kg/m2.
3. Subject has a diagnosis of uterine fibroids documented by a pelvic ultrasound.
4. Subject's menstrual cycles is between 21 days and 35 days in the last 3 months.
5. Subject has clinical manifestations of heavy menstrual bleeding.
6. Subject's menstrual blood loss >80mL for at least 2 menstrual periods assessed at screening using the alkaline hematin method.

Key Exclusion Criteria:

1. The subject is pregnant or breast-feeding or is planning a pregnancy within the duration of the treatment period of the study.
2. The subject has a history of uterus surgery that would interfere with the study.
3. The subject's condition is so severe that she will require surgery within 6 months.
4. The subject have had or are currently suffering from any estrogen- dependent malignancy.
5. The subject has a significant risk of osteoporosis, or have a known history of osteoporosis or other metabolic bone disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Responders based on menstrual blood loss (MBL) volume reduction at Week 24. | The last 28 days before the Week 24.
  MBL will be determined using the Alkaline Hematin method (AHM). Responder means whose MBL less than 80mL during the last 28 days before the Week 24 and more than 50% reduction in MBL compared to the baseline.

SECONDARY OUTCOMES:
Time to reduced MBL before the Week 24. | From baseline to Week 24.
  Reduced MBL means MBL less than 80ml and more than 50% reduction in MBL compared to the baseline.
Percentage of amenorrhea at the Week 24. | From baseline to Week 24.
  Amenorrhea is defined as having 0 data (or volume below the lower limit of quantification) from the AHM of MBL from the central laboratory or missing of AHM data with reported of "spotting" or "no bleeding" in the eDiary for 35 days before Week 24.
Time to amenorrhea before the Week 24. | From baseline to Week 24.
  The number of days from Study Day 1 to the first day having amenorrhea.
Days of menstrual bleeding in the last 28 days before the Week 24. | The last 28 days before the Week 24.
  Record the number of days.
Hemoglobin levels at the Week 24 in the subgroup of subjects with anemia. | The Week 24.
  Anemia is defined as hemoglobin below 12g/dL at baseline.

OTHER OUTCOMES:
Percentage of Responders at the Week 52. | The last 28 days before the Week 52.
  Responder is defined as above.
Time to reduced MBL before the Week 52. | From baseline to Week 52.
  Reduced MBL is defined as above.
Percentage of amenorrhea at the Week 52. | From baseline to Week 52.
  Amenorrhea is defined as above.
Time to amenorrhea before the Week 52. | From baseline to Week 52.
  The number of days from Study Day 1 to the first day having amenorrhea.
By 52 weeks, the number of days with menstrual bleeding per 28 days. | From baseline to Week 52.
  Record the number every 28days.
Score of Uterine Fibroids related pain, symptoms and quality of life. | From Week 12 to Week 64
  Use specified scales.
Bone Mineral Density (BMD) | The Week 24 and Week 52.
  Assessed by dual-energy X-ray absorptiometry (DXA) scan.
Adverse events | Up to Week 64.
  Clinical manifestation，frequency and severity of Treatment-Emergent Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Congjian Xu, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (29):
- China (29):
  - Site no.28, Beijing
  - Site no.31, Beijing
  - Site no.34, Beijing
  - Site no.11, Changchun
  - Site no.6, Changsha
  - Site no.7, Changsha
  - Site no.17, Chengdu
  - Site no.22, Chengdu
  - Site no.10, Chongqing
  - Site no.3, Guangzhou
  - Site no.4, Guangzhou
  - Site no.19, Hangzhou
  - Site no.21, Jinan
  - Site no.23, Lianyungang
  - Site no.14, Nanjing
  - Site no.15, Nanjing
  - Site no.16, Nanjing
  - Site no.26, Nanjing
  - Site no.18, Shanghai
  - Site no.1, Shanghai
  - Site no.29, Shanghai
  - Site no.8, Shenyang
  - Site no.30, Shenzhen
  - Site no.5, Taiyuan
  - Site no.2, Tianjin
  - Site no.20, Wenzhou
  - Site no.25, Wuhan
  - Site no.13, Xi'an
  - Site no.32, Zhengzhou

IPD SHARING:
Plan to Share IPD: No